CLINICAL TRIAL: NCT05539989
Title: Phase I/II Randomized, Placebo-Controlled Study of the Safety and Immunogenicity of VPM1002 Vaccination or BCG Revaccination Against Tuberculosis in Pre-Adolescents Living With and Without HIV in South Africa
Brief Title: Safety and Immunogenicity of VPM1002 Vaccination or BCG Revaccination Against TB in Pre-Adolescents Living With and Without HIV in South Africa
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study is no longer moving forward due to the changing TB vaccine landscape.
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMPAACT 2035/HVTN 604; UM1AI068632 (NIH); UM1AI068616 (NIH); UM1AI106716 (NIH); HHSN275201800001I (Other Grant/Funding Number: NICHD)
Record Dates: First submitted 2022-09-09; First posted 2022-09-14 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Tuberculosis; HIV Infections
Keywords: Bacterial and fungal diseases; Tuberculosis; Vaccine; Live vaccine; rBCG
MeSH Terms: conditions — Tuberculosis; HIV Infections; Mycoses | interventions — VPM1002 recombinant BCG vaccine; BCG Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VPM1002 Vaccine Arm (Experimental): Participants stratified by HIV and M.tb sensitization status.
  Interventions: Biological: VPM1002 Vaccine
- BCG Vaccine Arm (Experimental): Participants stratified by HIV and M.tb sensitization status.
  Interventions: Biological: BCG Vaccine
- Placebo Arm (Placebo Comparator): Participants stratified by HIV and M.tb sensitization status.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: VPM1002 Vaccine — 0.1 mL (2-8x10^5 CFU)
  Arms: VPM1002 Vaccine Arm
Biological: BCG Vaccine — 0.1mL (0.075 Mycobacterium bovis)
  Arms: BCG Vaccine Arm
Drug: Placebo — 0.1 mL (sodium chloride for injection 0.9%)
  Arms: Placebo Arm

SUMMARY:
The purpose of this study is to assess whether Mycobacterium bovis rBCGΔureC::hly (VPM1002) vaccination and Mycobacterium bovis bacille Calmette-Guérin (BCG) revaccination are safe and immunogenic in pre-adolescents with and without HIV and with and without Mycobacterium tuberculosis (M.tb) sensitization.

DETAILED DESCRIPTION:
Phase I/II, double-blinded, placebo-controlled, randomized (1:1:1) multi-center study. Randomization will be stratified by HIV status and M.tb sensitization status. The study will enroll approximately 480 pre-adolescents (8-14 years of age inclusive) with or without HIV and with or without M.tb sensitization who received BCG vaccination at birth. Participants with HIV will be immunocompetent and virologically suppressed on antiretroviral therapy.

Participants will be randomized to one of three study product arms: VPM1002 Vaccine, BCG Vaccine, or Placebo. Each participant will receive a single intradermal injection of the assigned study product.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian is willing and able to provide written informed consent; when applicable potential participant is willing and able to provide written assent
* Age 8-14 years (inclusive) at entry
* Received birth dose of BCG vaccine
* Has a negative nucleic acid test result for M.tb at screening and no other evidence of current active TB disease at screening
* M.tb sensitization status (positive or negative) determined based on IGRA testing at screening
* HIV status determined
* For participants living with HIV: has been receiving antiretroviral therapy for at least six months prior to study entry, has a CD4+ cell count of at least 200 cells/mm^3 at screening, has had a suppressed HIV viral load for at least three months prior to entry
* Has normal or grade 1 results for all of the following at screening: Hemoglobin, White blood cell count, Platelet count, Creatinine, ALT, AST, Total bilirubin
* Has a normal temperature and no signs or symptoms of acute illness
* For participants assigned female sex at birth or who could otherwise become pregnant: not pregnant
* For participants assigned female sex at birth or who could otherwise breastfeed: not breastfeeding
* Expected to be available for 48 weeks of study participation
* Not expected to participate in any other study of an investigational agent during the 48 weeks of study participation

Exclusion Criteria:

* Known significant exposure to TB or receipt of tuberculin skin test in the six months prior to study entry
* Receipt of treatment for active TB disease in the 24 months prior to study entry
* Receipt of TB preventive therapy within 30 days prior to study entry or expected to initiate TB preventive therapy within the 48 weeks following study entry
* For participants living with HIV, current active AIDS-defining condition
* Receipt of any of the following: Any investigational TB vaccine, More than 14 consecutive days of systemic immunosuppressants or other immune-modifying therapy within the six months prior to study entry, Any immunoglobulin or other blood product within the three months prior to study entry,
* Receipt of any vaccine within the 30 days prior to study entry or is expected to receive any vaccine between study entry and the Week 4 Visit
* Receipt of allergy treatment with an antigen injection within the 30 days prior to study entry or is expected to receive one or more antigen injections between study entry and the Week 48 Visit
* History of any of the following: serious adverse reaction to any vaccine, allergy or hypersensitivity to BCG vaccine, allergy or hypersensitivity to the components of VPM1002 vaccine, anaphylaxis, generalized urticaria, autoimmune disease, diabetes mellitus type 1 or type 2, mild persistent, moderate, or severe asthma, bleeding disorder, malignancy, any condition resulting in the absence of a functional spleen (asplenia), including but not limited to sickle cell disease
* History of seizure or use of any medication to prevent or treat seizure within the three years prior to entry
* History of suspected or confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection diagnosed within the 30 days prior to entry
* Any other documented or suspected clinically significant medical, psychiatric, or behavioral condition or any other condition that, in the opinion of the site investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
All adverse events | Through Week 48
  Proportion of participants, based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017
Solicited adverse events | Through Week 16
  Proportion of participants, based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017
Grade 3 or higher adverse events | Through Week 48
  Proportion of participants, based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017
Serious adverse events | Through Week 48
  Proportion of participants, based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017
Adverse pregnancy outcomes | Through Week 48 or delivery or other pregnancy outcome, whichever occurs later
  Proportion of participants, based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017
Frequency and response of VPM1002-specific and BCG-specific CD4+ and CD8+ T cells expressing Th1 and/or Th17 cytokines | Through Week 10
  Measured by ICS and flow cytometry on cryopreserved PBMCs

SECONDARY OUTCOMES:
Frequency and response of VPM1002-specific and BCG-specific CD4+ and CD8+ T cells expressing Th1 and/or Th17 cytokines | Weeks 24 and 48
  Measured by ICS and flow cytometry on cryopreserved PBMC
Mycobacteria-specific IgA, IgG, and IgM binding antibodies | Entry and Weeks 4, 10, 24, and 48
  Measured using BAMA
Association of HIV and IGRA with primary safety outcomes (All AEs, solicitated AEs, grade 3 or higher AEs, serious adverse events, adverse pregnancy outcomes). | Through Week 48 or delivery or other pregnancy outcome, whichever occurs later
  Based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017
Cellular immunogenicity outcome measures associated with HIV and IGRA status | Through Week 48
  VPM1002-specific and BCG-specific CD4+ and CD8+ T cells expressing Th1 and/or Th17 cytokines, measured by ICS and flow cytometry on cryopreserved PBMCs
Humoral immunogenicity outcome measures associated with HIV and IGRA status | Through Week 48
  Mycobacteria-specific IgA, IgG, and IgM binding antibodies, measured using BAMA
Gene expression profiles | Entry and Weeks 1, 4, and 10
  Measured by RNA-seq in whole blood
Differential leukocyte count and immunophenotype | Entry and Weeks 1, 4, and 10
  Measured in cryopreserved ex vivo whole blood (DLC-ICE) by flow cytometry
Measurement of soluble proinflammatory mediators | Entry and Weeks 1, 4, and 10
  Based on serum measurement
Acceptability of the study products | Week 24
  Based on scores derived from questionnaire responses

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Marie Cranmer, MD, MPH, Study Chair — Emory University
Locations (9):
- South Africa (9):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Setshaba Research Centre CRS, Soshanguve, Gauteng
  - Isipingo CRS, Soshanguve, KwaZulu-Natal
  - Klerksdorp CRS, Klerksdorp, North West
  - Desmond Tutu TB Centre - Stellenbosch University (SU) CRS, Cape Town, Western Cape
  - Emavundleni CRS, Cape Town, Western Cape
  - Umlazi CRS, Durban
  - Wits RHI Shandukani Research CRS, Johannesburg
  - Family Clinical Research Unit (FAM-CRU) CRS, Tygerberg Hills

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses? To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available?
  Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/studies/submit-research-proposal. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.
URL: https://www.impaactnetwork.org/studies/submit-research-proposal